CLINICAL TRIAL: NCT01537367
Title: Intervention Trials to Retain HIV-positive Patients in Medical Care
Brief Title: Intervention to Retain HIV-positive Patients in Medical Care
Acronym: Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CDCHRSA9272007
Record Dates: First submitted 2012-02-10; First posted 2012-02-23 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Primary Care Appointment Keeping
Keywords: Human immunodeficiency virus; HIV primary care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enhanced contact only (Experimental): Patients allocated to the Enhanced contact only arm will receive:
  HIV information and education
  * Specific to importance of coming to care regularly
  * Generic and tailored components
  * Approximately 10 minutes in length
  Enhanced contact over time
  * Collect locator information
  * Follow-up contact after medical visit (face-to-face or phone)
  * Appointment reminders (telephone, e-mail, text message)
  * Periodic telephone contact across time (support, update locator info, refer any unmet needs to Case Manager)
  * Attempt to make immediate contact following a missed visit and re-schedule appointment (use locator contact info)
  Interventions: Behavioral: Enhanced contact only
- Enhanced contact plus behavioral skills (Experimental): Enhanced contact plus behavioral skills is the longer experimental intervention arm.
  Interventions: Behavioral: Enhanced contact plus behavioral skills
- Standard of Care (Active Comparator): Patients assigned to control arm will receive the standard services offered to all patients at the clinic.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Enhanced contact plus behavioral skills — The enhanced contact plus behavioral skills arm is the longer experimental arm.
  Arms: Enhanced contact plus behavioral skills
Behavioral: Enhanced contact only — The enhanced contact only arm is the shorter experimental arm.
  Arms: Enhanced contact only
Behavioral: Standard of Care — The standard of care arm is the comparison group arm that receives only standard clinical services.
  Arms: Standard of Care

SUMMARY:
PROJECT OVERVIEW

This research is a collaboration between the Centers for Disease Control and Prevention (CDC), the Health Resources and Services Administration (HRSA), and six university-affiliated HIV clinics in the United States.

Study title: Intervention Trials to Retain HIV Patients in Medical Care

Study sites: The study will be performed at six HIV clinics affiliated with academic medical centers.

Objectives: Using HIV patients' clinical data (without personal identifiers) routinely archived in electronic databases at the six participating clinics do the following:

• To examine the extent to which a client-centered intervention delivered by trained interventionists (Phase 2 trial of the project) improves patient attendance for HIV primary care over and above the effect of the clinic-wide intervention. Phase 2 is a three-arm randomized controlled trial conducted at each of the participating six clinics. 300 patients will be enrolled in the Phase 2 trial at each clinic. One hundred will be new patients and 200 will be patients with inconsistent attendance for HIV primary care at the clinic in the prior 12 months. Patients will be randomized to: (1) an enhanced contact plus behavioral skills arm or (2) an enhanced contact-only arm in which patients will receive a longer or a shorter client-centered intervention from two trained interventionists, or (3) the standard of care arm in which patients will receive the clinic-wide intervention and routine HIV clinical care only.

DETAILED DESCRIPTION:
Design: Phase 1 uses a pre-post comparison of clinic attendance rates before and during a clinic-wide intervention. Phase 2 uses a randomized controlled trial experimental design.

Target population: Adults in primary medical care for HIV infection at 6 sites: (1) University of Alabama at Birmingham; (2) Baylor College of Medicine, Houston, Texas; (3) Johns Hopkins University School of Medicine, Baltimore, Maryland; (4) State University of New York, Downstate Medical Center, Brooklyn, New York; (5) Boston Medical Center, Boston, Massachusetts; and (6) University of Miami Miller School of Medicine, Miami, Florida.

Primary endpoints: The proportion of patients attending one or more HIV primary care visits in each of three four-month periods over the 12-months. A second measure will be the percentage of kept divided by scheduled primary care visits, excluding cancelled visits.

Duration of study: In the Phase 2 trial, the enrollment period will run six months and the three-arm intervention will run 12 months.

Main eligibility criteria: Phase 1: All patients presenting at the clinics beginning April 1, 2009 will receive the clinic-wide intervention. Attendance data from electronic medical records will be archived at the clinics (and transmitted later to CDC) beginning on April 1, 2008, one year before the start of the clinic-wide intervention. Patients with at least one scheduled clinic appointment qualify for inclusion in the study database. In Phase 2, patients 18 years of age and older (19 years of age in Alabama) who meet one of the following criteria are eligible to enroll: (1) new patients (first or second care visit at the clinic), or (2) patients who have inconsistent attendance for HIV primary care--defined as having had at least one no-show for a primary care appointment in the prior 12 months and patients not seen for HIV primary care at least once in each of two consecutive 6-month periods (among persons who have been patients at the clinic for at least 12 months.)

Study procedures: In Phase 1, attendance data maintained in electronic databases at the six participating clinics will be used (without personal identifiers) to examine attendance rates before and during the clinic-wide intervention. The Phase 1 clinic-wide intervention will include hanging posters in the clinic and having clinic staff distribute brochures that address the importance of attending HIV care on a regular basis, the importance of re-scheduling and canceling appointments, and having HIV primary care providers deliver brief messages about the importance of regular clinic attendance to all patients.

In Phase 2 trial, eligible patients (determined by review of attendance data from the clinic's database) will be consented, enrolled, and randomized to receive either (1) an enhanced contact plus skills intervention or (2) an enhanced contact only intervention from two trained interventionists, or (3) to receive standard of care at the clinic (no contact with the interventionists). The Phase 2 trial intervention includes periodic one-on-one meetings with the interventionists to address barriers to care (attitudes about HIV and unmet needs such as transportation, child care, housing, mental health, and drug use). The interventionists will work in collaboration with the patient's existing case manager(s) to help address these needs. Additionally, the interventionists will develop a personalized retention plan based on the patient's responses to a retention risk screener, deliver information and motivational statements about the importance of regular medical care for HIV infection, help the patient learn how to navigate a complex medical system, maintain contact (e.g., via telephone or outreach visits) with patients between clinic appointments, and make reminder telephone calls a few days before appointments.

Attendance data:

Enrollees' HIV primary care clinic attendance will be monitored quarterly through electronic medical records for at least 18 months, six months before and 12 months during the intervention. Patients who are not enrolled in the trial will continue to receive regular medical care at the clinic as well as the clinic-wide intervention.

Analysis methods: In Phase 1, a cohort of patients at each clinic will be identified and followed over time to compare their attendance (through electronic medical records) before and during the clinic-wide intervention using appropriate methods for making pre-post comparisons. In the Phase 2 trial, attendance will be compared by intervention arm and further broken down by demographic (e.g., gender, race/ethnicity) and clinical subgroups (e.g., viral load at baseline, self-reported substance use) to examine variables that may modify the intervention effect.

Data Management:

Data management and analysis will be the primary responsibility of CDC, although sites will also participate in data analysis activities. CDC will train sites in data management and in the use of the Secure Data Network (SDN) to transmit data files to CDC. CDC will provide all necessary data management guidelines to research sites.

Protocol Development:

CDC and HRSA will have the lead responsibility for the development of the project protocol for local IRB review by all cooperating institutions participating in the research project. HRSA in collaboration with CDC, will organize and conduct site investigators' meetings to discuss the project's progress and plan for the next year's milestones.

Protocol Modifications:

All protocol modifications will be approved by local site IRBs. Local IRB approvals will be obtained before protocol changes are implemented. CDC will maintain copies of current local site IRB approval letters and approved consent forms.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet ONE of the following three clinic attendance criteria:

  * Intake visit or 1st or 2nd HIV primary care visit at the clinic
  * At least one no-show for an HIV primary care appointment in the prior 12 months (includes patients who may not have had a full 12-month history at the clinic)
  * Not seen for HIV primary care at least once in each of two consecutive 6-month periods (among patients who have been seen at the clinic for at least 12 months)
* In addition, patients must meet ALL of the following personal criteria:

  * 18 year of age or older (at least 19 years of age in Alabama)
  * An HIV-positive patient receiving care at the clinic
  * Able to speak English or Spanish
  * No plans to move out of the area in the next 12 months
  * Able to provide informed consent

Exclusion Criteria:

* Failure to meet one of the three attendance criteria or failure to meet all of the personal criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1838 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lytt Gardner, Ph.D., Study Director — Centers for Disease Control and Prevention, Division of HIV/AIDS Prevention
Locations (6):
- United States (6):
  - 1917 Clinic of the University of Alabama-Birmingham, Birmingham, Alabama
  - Adult HIV Clinic of the Jackson Health System, Miami, Florida
  - Moore Clinic of the Johns Hopkins University Medical Institutions, Baltimore, Maryland
  - Boston University Medical Center, HIV Clinic, Boston, Massachusetts
  - SUNY Downstate Medical Center, STAR Health Center, Brooklyn, New York
  - Baylor College of Medicine-Thomas Street Health Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from June 15, 2010 through February 11, 2011. Recruitment time varied from 6 months to 8 months, by clinic site. Recruitment always occurred during regularly scheduled primary care appointments, either in a private corner of the waiting room, or in an adjacent room of the clinic.
Pre-assignment Details: No exclusions from the trial if participant was deemed eligible and agreed to participate. Once participants were deemed eligible, and agreed, they were escorted to a private room to do the audio-CASI questionnaire. After the audio-CASI was completed they were immediately randomized to one of the three arms.
Groups:
- Enhanced Contact-only: The enhanced contact only arm was described in the summary/Detailed Description as the shorter intervention. This arm did not require any additional special study visits after enrollment. The contacts of the interventionist with the patient were related to making and keeping clinic appointments.
- Enhanced Contact-plus Behavioral Skills: This arm was described in the summary/Detailed Description as the "longer comprehensive intervention arm". Patients assigned to this arm were required to return to the clinic within the next two weeks after enrollment to receive a one-to-two hour training in elements of behavioral skills relevant to improved clinic attendance. The mixture of elements was determined by the interventionist in a discussion with the patient at this special study visit. Subsequent contacts of the interventionist with patients in this arm would refer to these behavioral skills elements and to making and keeping clinic appointments.
- Standard of Care: Participants randomized to the SOC arm received the usual attention and encouragement to attend all clinic visits that prevailed at the clinic at the time of this intervention. This attention could include the routine advice from a nurse, personal or robo reminder calls before a next clinic visit. Contacts with case managers and social workers related to clinic appointments could also occur, per the clinic's standard procedures.
Period: Overall Study
Arm/Group | Enhanced Contact-only | Enhanced Contact-plus Behavioral Skills | Standard of Care
Started | 615 | 610 | 613
Completed | 615 (All participants who were enrolled were followed for routine HIV clinic attendance via clinic EMR.) | 610 (All participants who were enrolled were followed for routine HIV clinic attendance via clinic EMR.) | 613 (All participants who were enrolled were followed for routine HIV clinic attendance via clinic EMR.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The transgendered particpants were all males at birth, so we added the transgendered to the male count in the gender field.
Groups:
- Enhanced Contact-only: The enhanced contact only arm was described in the summary/Detailed Description as the shorter intervention. This arm did not require any additional special study visits after enrollment. The contacts of the interventionist with the patient related to making and seeing clinic appointments.
- Total: Total of all reporting groups
Arm/Group | Enhanced Contact-only | Enhanced Contact-plus Behavioral Skills | Standard of Care | Total
Number analyzed (Participants) | 615 | 610 | 613 | 1838
Age, Customized [Number; unit: participants] — Five-category Age Age groups: 18-29 30-39 40-49 50-59 60-plus
  participants
    18-29 years | 59 | 67 | 73 | 199
    30-39 years | 118 | 121 | 122 | 361
    40-49 years | 210 | 202 | 212 | 624
    50-59 years | 187 | 176 | 167 | 530
    60-plus years | 41 | 44 | 39 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 234 | 228 | 665
  Male | 412 | 376 | 385 | 1173
Race/Ethnicity, Customized [Number; unit: participants] — Mutually exclusive categories where Hispanic is treated as a distinct race category, over-riding any other selection from the OMB race variable.
  participants
    Black | 431 | 422 | 409 | 1262
    White | 87 | 72 | 76 | 235
    Other race | 18 | 15 | 20 | 53
    Hispanic | 79 | 101 | 108 | 288

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Attending a Primary Care Visit in Each of 3 Four-month Periods (First Measure)
Description: Kept visits for each patient were assessed in 4-month periods over the 12 months of the intervention. This is a binary measure, requiring attendance at least once in each of the three 4-month periods.
Time Frame: 12 months after enrollment
Population: Intention to Treat (ITT)
Measure: Number; unit: percent in care each 4 month period
Arm/Group | Enhanced Contact-only | Enhanced Contact-plus Behavioral Skills | Standard of Care
Number analyzed (Participants) | 615 | 610 | 613
percent in care each 4 month period | 55.8 | 55.6 | 45.7

2. Secondary Outcome: Mean Counts Per Person (Rates) of Kept Visits.
Description: The rate of kept clinic visits per person over 12 months.
Time Frame: 12 months after enrollment
Measure: Mean (Standard Error); unit: # kept visits/person/12 months
Arm/Group | Enhanced Contact-only | Enhanced Contact-plus Behavioral Skills | Standard of Care
Number analyzed (Participants) | 615 | 610 | 613
# kept visits/person/12 months | 4.12 (0.118) | 4.15 (0.115) | 3.59 (0.096)

3. Primary Outcome: The Percentage of Kept Divided by Scheduled Primary Care Visits, Excluding Cancelled (Second Measure).
Description: Primary care visits are scheduled appointments for HIV-positive patients to see a physician, nurse practitioner, or physician assistant (a provider who can prescribe medication) at the HIV clinic.
Time Frame: 12 months after enrollment
Population: Intention to Treat (ITT)
Measure: Number; unit: Percentage of Pt kept visits/#scheduled
Arm/Group | Enhanced Contact-only | Enhanced Contact-plus Behavioral Skills | Standard of Care
Number analyzed (Participants) | 615 | 610 | 613
Percentage of Pt kept visits/#scheduled | 72.5 | 70.9 | 67.2

ADVERSE EVENTS:
Arm/Group | Enhanced Contact-only | Enhanced Contact-plus Behavioral Skills | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/615 | 0/610 | 0/613
Other Adverse Events (participants affected / at risk) | 0/615 | 0/610 | 0/613

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No